CLINICAL TRIAL: NCT04362462
Title: Genomic/Molecular Profiling of Residual Disease After Neoadjuvant Chemotherapy in Hispanic/ Latino Women With Triple-negative Breast Cancer
Brief Title: Molecular Profiling After Neoadjuvant Chemotherapy for Triple-negative Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Alexander Philipovskiy, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E19059
Record Dates: First submitted 2019-12-18; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — breast cancer tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neoadjuvant chemotherapy (NACT) can induce complete pathologic response (pCR) in approximately 35-55% of patient with triple-negative breast cancer (TNBC). These patients have excellent long term survivals. On the other hand patients with residual disease exhibit a high rate of local or metastatic. Although it has been successful in some regards, randomized trials have shown similar rates of mortality between patients receiving NACT and adjuvant chemotherapy (ACT). The goal of this study is to understand the molecular biology (gene expression signature) driving treatment-resistant TNBC. The investigators are planning to identify targetable genetic alterations which may help to optimize adjuvant therapy for the patient with residual TNBC.

DETAILED DESCRIPTION:
In this study, investigators will understand the clinical relevance of genomic heterogeneity of triple-negative breast cancer by determining pathological complete response (pCR) rates after NACT, based on genomic profiling of individual tumors. Investigators will identify new genomic alterations in patients with residual TNBC as well as in patients who develop metastatic disease within 24 months after completion of all appropriate therapies. Investigators will demonstrate unique genomic alteration, and we will identify new tumor markers in Hispanic/Latino (H/L) women with TNBC.

Inclusion Criteria:

This study aims to include all patients with early stage (I-III) TNBC who received NACT and subsequently underwent surgical treatment (mastectomy or lumpectomy) or women with triple-negative breast cancer who progressed and developed metastatic disease within 24 months after all appropriate therapies.

1. Age > 18 or <86 years of age, for Hispanic/Latino women we will use the National Advisory Committee on Racial, Ethnic and Other populations NAC definition which is (the ethnonyms "Hispanic" and "Latino" to refer collectively to the inhabitants of the United States of America who are of Latin American or Spanish origin-that is, Latino or Hispanic Americans).
2. Pre- and Post - menopausal women with histologically confirmed hormonal receptor negative (ER and/or PR <1%), Her2-neu - negative (by IHC or/and FISH) invasive breast cancer stages I - III or with metastatic triple-negative breast cancer (if develop metastatic disease during the chemotherapy or within 24 months after completion of all appropriate treatments).
3. Patients must be eligible for NACT, and surgical lumpectomy or mastectomy.
4. All patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with Institutional and Federal guidelines.

Exclusion Criteria:

1. Women < 18 or >86 years of age
2. ER/PR- positive, Her-2 neu - positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 or <86 years of age, for Hispanic/Latino women we will use the National Advisory Committee on Racial, Ethnic and Other populations NAC definition which is (the ethnonyms "Hispanic" and "Latino" to refer collectively to the inhabitants of the United States of America who are of Latin American or Spanish origin-that is, Latino or Hispanic Americans).
2. Pre- and Post - menopausal women with histologically confirmed hormonal receptor negative (ER and/or PR <1%), Her2-neu - negative (by IHC or/and FISH) invasive breast cancer stages I - III or with metastatic triple-negative breast cancer (if develop metastatic disease during the chemotherapy or within 24 months after completion of all appropriate treatments).
3. Patient must be eligible for neo-adjuvant chemotherapy, and surgical lumpectomy or mastectomy.
4. All patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with Institutional and Federal guidelines.

Exclusion Criteria:

1. Women < 18 or >86 years of age
2. ER/PR- positive, Her-2 neu - positive breast cancer.

Ages: 18 Years to 86 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The majority of triple-negative breast cancer patients are female.
Study Population: Females with confirmed triple-negative breast cancer.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 12-24 months
  Progression free survival at one and two years in order to avoid unnecessary chemotherapy in patients with chemotherapy resistant tumors. We will measure and track the response rate to chemotherapy as well as pathological complete response after chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Philipovskiy, MD, PhD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech University Health Sciences Center- El Paso, El Paso, Texas, United States